CLINICAL TRIAL: NCT04635410
Title: Ultrasound Prediction of Delivery Mode: Can the First Stage Prediction Model be Further Improved?
Brief Title: Improving Ultrasound Based Prediction of Delivery Mode
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 283692
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: NO CONDITIONS
Keywords: NO CONDITIONS
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ULTRASOUND IMAGING — SCAN LABOURING WOMEN BY ULTRASOUND

SUMMARY:
The progress of labour is traditionally determined by regular vaginal examinations (VEs) to assess the cervix (neck of the womb) and the baby's head position. Such examinations can be uncomfortable and risk causing infection to the baby or mother's womb. The findings are subjective, can be unreliable and cannot be recorded for later review and analysis.

The novel, non-intrusive "transperineal ultrasound" technique has been developed utilising existing scanning machines normally found on a delivery unit, with the ultrasound probe placed outside the woman's vagina. This allows objective, recordable measurements creating images that can be captured and stored electronically.

This is a prospective longitudinal observational cohort study in nulliparous term (37-42 weeks) labouring women. This study aims to improve the prediction of intrapartum Caesarean Delivery (ICD).

The study contains ultrasound and clinical assessments:

Transabdominal Ultrasound to measure: Umbilical and Middle Cerebral Artery Doppler, fetal head position and Amniotic Fluid Index (AFI).

Transperineal Ultrasound to assess: Head Perineum Distance (HPD), Caput Succedaneum and moulding.

Digital vaginal examination by a caregiver: to measure cervical dilatation.

Primary outcome:

• Mode of delivery

Secondary outcome:

• Time to delivery

Neonatal outcomes:

• Apgar score, cord pH level, gender, fetal birth weight, neonatal unit admission within 24 hours, neonatal morbidity.

DETAILED DESCRIPTION:
Intrapartum Caesarean Delivery (ICD) in advanced labour has a greater fetal and maternal morbidity and mortality than an elective prelabour Caesarean delivery. The prediction of delivery mode may reduce the likelihood of intrapartum Caesarean delivery. There is also a parental desire to know the likelihood of vaginal delivery. Women admitted to delivery units throughout the world undergo internal digital vaginal examination (DVE) when they are thought to be in labour or where a diagnosis of labour needs to be discounted. DVE is an uncomfortable experience, multiple examinations have been linked to ascending maternal and fetal infection, and it is subjective method and not reliable technique to assess labour progress.

It has recently become possible to make assessments more objectively using ultrasound. Ultrasound in labour (intrapartum ultrasound) has come to the forefront in the last decade stemming from a persistent demand for a more reliable method of labour assessment coupled with a wider availability of ultrasound on the delivery suite.

The hypothesise in this study, that developing the previously derived proof of principle labour prediction model for nulliparous women and using an additional data could improve the prediction accuracy of intrapartum Caesarean delivery by developing a robust model.

Using the additional data gathered in term nulliparous patients, will develop the model to predict pregnancy outcomes. This may aid in delivery of care to pregnant women by providing a real-time online calculation tool for the likelihood of Caesarean delivery and length of labour based on repeat ultrasound measurements.

All participants will be identified by the researcher and an emphasis will be placed on recruiting patients antenatally as much as possible. All participating patients will be consented prior to enrolment and will receive a full explanatory information leaflet. If recruited antenatally, there is no time limit until the woman enters the delivery unit. If recruited in labour, then 2 hours will be considered appropriate to make a decision on whether they wish to take part and patient will only be approached when relatively pain-free (in between contractions).

The admission ultrasound scan will include if feasible fetal Doppler assessment of the Umbilical Artery (Umb A) and Middle Cerebral Artery (MCA). Amniotic Fluid Index (AFI) will also be measured. The fetal position will be assessed with a transabdominal scan and recorded.

Firstly, Umb A and MCA Doppler in addition to the fetal position and AFI, will be assessed with a transabdominal scan. After that, the transducer will be placed transperineally at the level of the posterior fourchette in a transverse position to measure HPD while caput succedaneum will be measured in a sagittal transperineal scan. The moulding will be assessed as either present or not.

During the ultrasound examination, women will be in the supine position with flexed hips and knees and the bladder empty as previously described. Healthcare professionals will be blinded to the ultrasound findings, and these findings will also not be disclosed to the parents. Another doctor or midwife will perform all the ultrasound examinations. Subsequent scans will be performed as required at the time of routine clinical examinations typically between 2-4 hours apart but it may be longer.

The healthcare professional will perform DVE for assessment of cervical dilatation in line with the National Institute of Health and Clinical Excellence (NICE) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-44.
* Cephalic presentation.
* Nulliparous.
* Singleton.

Exclusion Criteria:

* Younger than 18 years.
* Life-threatening maternal or fetal compromise needing immediate medical attention and/or delivery.
* Women who in the opinion of the researcher are unable to give fully informed consent to the study.
* Non-cephalic presentations.
* Multiple pregnancies.
* Multiparous patients.
* Not in established labour

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — LABOURING WOMEN
Study Population: Recruitment will start upon approval of the study. The infrastructure, research fellow, ultrasound machines, and the database are already in place, which ensure that the study can start promptly upon approval, without affecting or compromising routine clinical service provision. We aim to recruit minimum number according to the following calculations:
  In the labour prediction model, there are approximately 12 variables with 10 patients needed per variable and an approximate 25% Caesarean section rate (the primary outcome) in the UK currently.
  Practical calculation:
  12 x 10 x (100/25) = 480 patients
  For predictive modelling, 480 patients minimum are required (37- 42 weeks). We have recruited 269 patients in the previous study, therefore, approximately 211 fully evaluable patients will be needed. We intend to recruit 240 participants to allow approximately 10% incomplete data/study withdrawals
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Intrapartum Caesarean delivery (ICD) | 3 years
  Number of participants who delivered by Caesarean section

SECONDARY OUTCOMES:
Time to delivery (length of labour of onset of the first stage to the completion of the second stage). | 12-24 hours
  Number of hours from the onset of labour to the end of the second stage

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial college NHS Trust Queen Charlotte and Chelsea Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided